CLINICAL TRIAL: NCT02356107
Title: 5-hydroxytryptophan and Creatine for Treatment Resistant Depression Associated With Hypoxia in Females
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Perry Renshaw (Other)
Responsible Party: Sponsor-Investigator, Perry Renshaw, MD, PhD, MBA, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5HTP/Creatine
Record Dates: First submitted 2015-01-27; First posted 2015-02-05 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 5-Hydroxytryptophan; Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label treatment with 5-HTP and Creatine (Experimental)
  Interventions: Drug: 5-hydroxytryptophan and Creatine monohydrate

INTERVENTIONS:
Drug: 5-hydroxytryptophan and Creatine monohydrate

SUMMARY:
The investigators hypothesize that the administration of two widely available, naturally occurring dietary supplements, 5 hydroxytryptophan and creatine monohydrate, will reduce the severity of depression in individuals exposed to chronic hypoxia by living at altitude. The purpose of this study is to determine if 8 weeks of dietary augmentation with oral 5 g creatine daily and 100 mg 5-HTP twice daily reduces hypoxia-related depressive symptoms measured by the 17-item Hamilton Depression Rating Scale (HAM-D) in women with SSRI or SNRI-resistant depression.

DETAILED DESCRIPTION:
Serotonin and creatine are processed separately in the brain, and deficits in these brain biochemicals lead to distinct clinical problems. Therefore, investigators believe that treatment with a combination therapy, which could correct both deficits, would have a synergistic effect in the treatment of hypoxia-related depression and possibly other forms of treatment-resistant depression. Thus, investigators propose to investigate antidepressant efficacy of dietary 5-hydroxytryptophan (5-HTP) and creatine, as a means to restore the brain neurotransmitter and metabolic imbalances linked to chronic hypoxia caused by high altitude residence.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, ages 18-64 years inclusive
* Current diagnosis of Major Depressive Disorder identified by the SCID-5-CT
* Current HAM-D17 score of > 15
* Adequate adherence to any FDA approved SSRI or SNRI for at least 8 weeks

Exclusion Criteria:

* Diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder, identified by the SCID-5-CT
* History of or current diagnosis of renal disease, such as chronic renal failure, acute renal failure or end stage renal disease
* Diabetes type I or II
* Colitis or diverticulitis
* History of pulmonary disease
* History of fibromyalgia, lupus, eosinophilia myalgia syndrome, dermatomyositis, polymyositis, rheumatoid arthritis, psoriatic arthritis, mixed connective tissue disease, ankylosing spondylitis, or other related rheumatological condition
* Seizure disorder
* Current serious suicide risk identified by the Columbia Severity Suicide Rating Scale
* Current treatment with an antipsychotic, mood stabilizer, or non-SSRI antidepressant
* Positive pregnancy test
* Previous diagnosis of serotonin syndrome
* Use of any excluded drugs or medications including serotonergic drugs or medications

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry F. Renshaw, MD, PhD, MBA, Study Director — University of Utah
Locations (1):
- University of Utah/The Brain Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Treatment With 5-HTP and Creatine: 5-hydroxytryptophan and Creatine monohydrate
Period: Overall Study
Arm/Group | Open Label Treatment With 5-HTP and Creatine
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Treatment With 5-HTP and Creatine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale
Description: The purpose of this study is to determine if 8 weeks of dietary augmentation with oral 5 g creatine daily and 100 mg 5-HTP twice daily reduces hypoxia-related depressive symptoms measured by the 17-item Hamilton Depression Rating Scale (HAM-D) in women with SSRI or SNRI resistant depression. HAM-D (outcome measure) was used to assess the level of depression at baseline and after 8 weeks of using the study drug. The Hamilton Depression Rating Scale ranges from 0 to 50. A score of 0-7 is considered to be normal. A score of 8-13 indicates mild depression. A score of 14-18 indicates moderate depression. Scores higher than 19 indicate severe depression.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Treatment With 5-HTP and Creatine
Number analyzed (Participants) | 15
units on a scale
  Baseline | 18.9 (2.5)
  After 8 weeks of treatment | 7.5 (4.4)

ADVERSE EVENTS:
Arm/Group | Open Label Treatment With 5-HTP and Creatine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 7/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment With 5-HTP and Creatine (N=15)
cold/flu symptoms (General disorders) | 1 (1)
kidney stones (Renal and urinary disorders) | 1 (1)
diagnosis of medullary sponge kidney (Renal and urinary disorders) | 1 (1)
injury/fall (Injury, poisoning and procedural complications) | 2 (2)
night sweats/ increased sweating (Endocrine disorders) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No